CLINICAL TRIAL: NCT06556199
Title: The Efficiency and Safety of Selinexor in Combination With Temozolomide and Anti-PD-1 Antibody in Patients With Relapsed/Refractory Primary Central Nervous System Lymphoma: A Prospective, Single-arm, Open, Phase Ib/II Clinical Study
Brief Title: A Study of Selinexor in Combination With Temozolomide and Anti-PD-1 Antibody in Patients With Relapsed/Refractory Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R202333
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-08

CONDITIONS: Relapsed/Refractory Primary Central Nervous System Lymphoma
MeSH Terms: conditions — Recurrence | interventions — selinexor; Temozolomide; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- selinexor-based treatment (Experimental)
  Interventions: Drug: Selinexor; Drug: Temozolomide; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Selinexor — Selinexor dose escalation: 40,60,80mg respectively every week, and dose expansion at the RP2D of Selinexor,every 3 weeks for 6 cycles.
Drug: Temozolomide — Temozolomide 150mg/m2 po d1-5 every 3 weeks for 6 cycles.
Drug: Anti-PD-1 monoclonal antibody — The dose of anti-PD-1 monoclonal antibody is fixed dose 200 mg intravenously every 3 weeks until until disease progression or recurrence, intolerance of toxicity, death, loss of follow-up, withdrawal of notification (whatever happened first).

SUMMARY:
This study is a prospective, single-arm, open label, Phase Ib/II clinical study to evaluate the safety and efficacy of selinexor in combination with temozolomide and anti-PD-1 monoclonal antibody in patients with relapsed/refractory primary central nervous system lymphoma(PCNSL). Phase Ib used a "3+3" dose-climbing design to confirm the safety, maximum-tolerated dose (MTD,if any) and recommended phaseII dose (RP2D) of selinexor in combination with fixed dose of temozolomide and anti-PD-1 monoclonal antibody for 6 cycles. Phase II was a comprehensive evaluation of efficacy and safety. Subjects who achieved complete remission or partial remission were treated with anti-PD-1 monoclonal antibody maintenance therapy until disease progression or recurrence, intolerance of toxicity, death, loss of follow-up, withdrawal of notification (whatever happened first).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 (inclusive).
* Participants must be able to understand and be willing to sign a written informed consent document.
* Eastern Cooperative Oncology Group performance status 0 to 3.
* Life expectancy of ≥ 3 months (in the opinion of the investigator).
* Primary central nervous system lymphoma (PCNSL) of B-cell origin confirmed by pathology (histology or cytology)
* Measurable disease was defined as at least ≥1.0cm in short-diameter by enhanced MRI.
* Recurrent/refractory PCNSL: Must have received at least one systemic treatment with methotrexate-based treatment.
* Any non-hematological toxicity associated with previous treatment should return to grade 1 or normal (except hair loss according to NCI CTCAE version 5.0)
* Bone marrow and organ function meet the following criteria (no blood transfusion within 14 days prior to screening, no G-CSF, no medication correction) :

  1. Bone marrow function: absolute value of neutrophils ≥1.5×10^9/L, platelets ≥80×10^9/L, hemoglobin ≥80 g/L;
  2. Liver function: serum total bilirubin ≤1.5×ULN (≤3.0×ULN, if there is liver metastasis); Glutamic oxalic aminotransferase (AST) and glutamic pyruvic aminotransferase (ALT) ≤2.5×ULN (≤5.0×ULN, if there is liver metastasis);
  3. Coagulation function: International standardized ratio (INR) and activated partial thrombin time ≤1.5×ULN;
  4. Renal function: serum creatinine ≤1.5×ULN or estimated creatinine clearance ≥60 mL/min (male: Cr (ml/min) = (140-age) × body weight (kg) /72× serum creatinine concentration (mg/dl); Female: Cr (ml/min) = (140- age) × body weight (kg) /85× serum creatinine concentration (mg/dl)
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 6 months after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 6 months after the last dose.
* Can accept multiple MRI/CT and lumbar puncture examination.
* Swallowing oral tablets/capsules without difficulty.
* Good compliance, willing to follow the visit schedule, dosing schedule, laboratory examination and other test procedure.

Exclusion Criteria:

* Pathological diagnosis was T cell lymphoma.
* Anti-tumor therapy with chemotherapy, radiotherapy, immunotherapy or antibody drugs, or Chinese herbal medicine with anti-tumor indications, small-molecule targeted therapy within 2 weeks, monoclonal antibody-coupled drugs or cytotoxin therapy within 10 weeks, and autologous stem cell transplantation within 6 months before the first administration.
* Participation in another clinical study with an investigational product during the 4 weeks prior to the first day of study treatment.
* Patients who use systemic adrenal corticosteroids for more than 5 days within 14 days prior to medication or who need to take >10mg of dexamethasone or equivalent drugs daily to control CNS disease.
* Active concurrent malignancy requiring active therapy.
* Prior treatment with temozolomide or anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs within 6 months prior to initial administration
* Have uncontrolled or significant cardiovascular disease, including (but not limited to) : Any of the following: congestive heart failure (NYHA Class III or IV);myocardial infarction; unstable angina; or the presence of an arrhythmia requiring treatment at the time of screening with a left ventricular ejection fraction (LVEF) < 50% in the 6 months prior to initial dosing; Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, undefined cardiomyopathy); A clinically significant history of prolonged QTc, grade II type II atrioventricular block or grade III atrioventricular block, or QTc interphase (method F) > 470 msec (female) or > 480msec (male);Atrial fibrillation (EHRA grade ≥2b);Patients with unmanageable hypertension were deemed unsuitable for participation in the study.
* Uncontrolled infections or infections that require intravenous antibiotic treatment.
* Chronic hepatitis B carriers with active hepatitis B or C infection (hepatitis B: acute hepatitis B, untreated chronic hepatitis B virus infection, HBV-DNA≥ the detection limit of each center; Hepatitis C: HCV RNA positive) or syphilis. Notes: Non-active HBV surface antigen (HBsAg) carriers, subjects with active HBV infection and persistent anti-HBV inhibition (HBV DNA < each center detection limit), and subjects cured of HCV can be enrolled.
* Human immunodeficiency virus (HIV) infection
* Clinically significant gastrointestinal abnormalities that may affect drug intake, transport, or absorption (such as active gastrointestinal inflammation, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy or gastric banding surgery.
* Prior allogenic stem cell transplant.
* For female subjects, they are currently pregnant or breastfeeding.
* Allergy to the investigational drug or excipient.
* The patient has active mental illness, alcohol, drug or substance abuse.
* The presence of any life-threatening disease, medical condition, or organ system dysfunction that the investigator believes may affect the patient's safety or compliance with the study procedure.
* There are other conditions that the investigator considers inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose | Up to 21days
  To determine the recommended phase 2 dose for Selinexor.
Objective response rate (ORR) for Phase II study | 18 weeks
  The objective response rate (ORR) is defined as the proportion of patients with CR or PR at the end of induction treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years after enrollment
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | Up to 2 years after enrollment
  OS is defined as the duration of time from start of treatment to time of death.
Duration of response | Up to 2 years after enrollment
  The duration of overall response is measured from the time achieving ORR to time of progression, relapse or death, whichever occurs first.

OTHER OUTCOMES:
ctDNA mutation and mean ctDNA concentration in serum and cerebrospinal fluid | Up to 2 years after enrollment
  Types of ctDNA mutations and frequency are measured by next generation sequencing. The mean ctDNA concentration is the concentration of ctDNA expressed as mean tumor molecules /ml at specific time points.
The levels of cytokine concentration in serum and cerebrospinal fluid | Up to 2 years after enrollment
  The levels of cytokine will be analyzed by ELISA in all patients recruited at Baseline and specific time point. The cytokine profile includes IL-6, IL-10, TNF-α, IFN-γ, IL-2 and IL-4

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No